CLINICAL TRIAL: NCT05309226
Title: Cannabis Use in Pregnancy and Downstream Effects on Maternal and Infant Health (CUPiD): A Pilot Prospective Cohort Study
Brief Title: Cannabis Use in Pregnancy and Downstream Effects on Maternal and Infant Health
Acronym: CUPiD
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Kingston Health Sciences Centre (Other); Children's Hospital of Eastern Ontario Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CTO 3791
Record Dates: First submitted 2022-02-10; First posted 2022-04-04 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Cannabis Use; Marijuana Use
Keywords: perinatal; cannabis; pregnancy; marijuana
MeSH Terms: conditions — Marijuana Use; Marijuana Abuse | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Consenting participants will be asked to contribute biological samples.
  We will allow participants to choose the scope of sample collection at each time-point. Sampling will be coordinated alongside routine clinical collections where possible to minimize burden to participants.
  Samples will be collected at 5 timepoints throughout the study time period: in each trimester of pregnancy, at delivery and at 6-12 weeks postpartum. Maternal blood and urine will be collected at all visits. During the delivery admission, cord blood, cord tissue, placenta, meconium, and breastmilk will be collected. At the postpartum visit, baby urine and blood (dried blood spot) and breastmilk will be collected.
  Partners will not be asked to contribute biological samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Pregnant Cannabis User: Pregnant individuals who disclose cannabis use in pregnancy
  We will examine patterns of cannabis use including the type of cannabis used, amount and frequency of cannabis use during the perinatal and postpartum periods. If participant decides to stop using cannabis in pregnancy, they will not be excluded from the study.
  Interventions: Other: Cannabis use in pregnancy or cannabis exposure in utero
- Pregnant Cannabis Non-User: Pregnant individuals who report not using cannabis in pregnancy and who have not used cannabis products for at least 3-months prior to pregnancy.
- Offspring of Pregnant Cannabis User: Infants born to pregnant participants who disclose cannabis use in pregnancy
  Interventions: Other: Cannabis use in pregnancy or cannabis exposure in utero
- Offspring of Pregnant Cannabis Non-User: Infants born to pregnant participants who report no cannabis use in pregnancy
- Partners: Partners of pregnant participants enrolled in this study.

INTERVENTIONS:
Other: Cannabis use in pregnancy or cannabis exposure in utero — Cannabis-related product use in pregnancy. Cannabis-related products will include all forms (e.g., dry flower, edibles, extracts, etc.) and formats of consumption (e.g., joint, bong, capsule, tincture, etc.).
  Groups: Offspring of Pregnant Cannabis User; Pregnant Cannabis User

SUMMARY:
With perinatal cannabis use rising in Canada, robust data on short-term and long-term effects on newborns are urgently needed. However, past barriers to obtain robust data included limited sample sizes, low self-reporting and no account of postpartum exposures. Therefore, this study will be conducted as a feasibility pilot study to tease out limitations that were present in previous studies. This study will help us dictate how to conduct a larger prospective cohort study to answer any knowledge gaps currently in the field of perinatal cannabis use.

DETAILED DESCRIPTION:
Since Canadian legalization of cannabis in October 2018, reports of cannabis use have increased even among pregnant women/individuals. Previous work has identified that cannabis products known as cannabinoids, such as THC, CBD, cannabinol and their metabolic by-products cross the placenta and can enter the fetal bloodstream and distribute throughout the fetal tissues, including the brain associating to neurodevelopmental outcomes. However, these studies were limited by their sample size, based on self-reporting and did not account for postpartum exposures. Notably, the CUPiD study is a pilot study to assess the feasibility for a larger prospective study and address past limitations.

We will aim to recruit 50 participants who are currently using cannabis in pregnancy and 50 participants who are not using cannabis in pregnancy within 12 months from either the Ottawa Hospital or Kingston General Hospital. The participants will be recruited any time in pregnancy and will be followed up until 4 months postpartum. Within the study period, there will be extensive data collection through surveys, diaries and medical chart reviews as well as biological sampling of the mother/birthing parent and the baby (after delivery).

This work will address key issues such as recruitment rate, level of engagement, protocol compliance and appropriateness of sample size and timeframe. By piloting a pregnancy cohort from which robust data on cannabis practices can be gathered, this project will lay the foundation for downstream research in this area.

ELIGIBILITY:
MOTHER INFANT DYADS

Inclusion Criteria:

Exposed and unexposed pregnant women/individuals must meet all of the following inclusion criteria at the time of enrollment to be eligible:

* Capacity to provide informed consent and to comprehend and comply with the study requirements
* Planning to deliver at TOH or KGH, or The Ottawa Birth and Wellness Centre (affiliated with TOH)
* Be ≥ 16 years of age at the time of consent

Exposed group: pregnant women/individuals who are using any cannabis-related product in pregnancy at the time of enrollment, or have used cannabis-related products in the current pregnancy for any reason (including but not limited to recreational use, to ease nausea and vomiting, use for chronic pain management or other medical indications).

Unexposed group: pregnant women/individuals who are not using cannabis-related products in pregnancy, and who have not used any cannabis-related product for at least 3-months prior to pregnancy.

Exclusion Criteria:

* Women/Individuals who self-report non-prescription use of controlled and illegal drugs in their current pregnancy (i.e., benzodiazepines, cocaine and crack, fentanyl, heroin, ketamine, lysergic acid diethylamide, magic mushrooms, MDMA, methamphetamine, gamma hydroxybutyrate, opioids, phenylcyclohexyl piperidine, salvia) or report their use in the 3-months prior to pregnancy. (**Use of alcohol or tobacco products prior to pregnancy or during pregnancy will not be an exclusion criterion**)
* Women/Individuals who self-report prescription use of opioid medications including methadone, Subutex, buprenorphine, tramadol, oxycodone, hydrocodone, and hydromorphine in their current pregnancy, or report their use in the 3 months prior to pregnancy
* Surrogate or planning to give child up for adoption

PARTNERS 'Partner' will be broadly defined as any individual identified as such by an enrolled pregnant participant (any sex or gender, any status - marital, common-law, or otherwise). Thus, eligible partners must meet all of the following inclusion criteria at the time of enrollment:

* Pregnant partner is enrolled in the CUPiD cohort study
* Have capacity to provide informed consent and to comprehend and comply with the study requirements
* Be ≥ 16 years of age at the time of consent

There are no pre-defined exclusion criteria for partners.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The primary study population will consist of pregnant individuals who are or are not using cannabis in pregnancy, and their infants. Partners will be invited to participate in a one-time survey.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Appropriateness of eligibility criteria | Within first year
  Measured by the reasons for exclusion of screened subjects
Recruitment rate | Within first year
  Measured by the proportion of eligible cases and controls recruited into the cohort
Level of engagement | Within first year
  Measured by the proportion of recruited subjects contributing data and biospecimens at each time point
Protocol compliance | Within first year
  Measured by attrition rate (loss to follow-up or withdrawal of consent) of enrolled subjects
Appropriateness of sample size and time frame | Within first year
  Measured by the timeframe required to recruit target sample size

SECONDARY OUTCOMES:
Fetal and neonatal morbidity (preterm) | Throughout pregnancy until 6-12 weeks postpartum
  Rates of: Preterm Birth (<37 weeks' gestation; 34 to 36 weeks' gestation (late preterm);32 to 33 weeks' gestation; 28 to 31 weeks' gestation; <28 weeks' gestation (very preterm birth))
Fetal and neonatal morbidity (sga) | Throughout pregnancy until 6-12 weeks postpartum
  Rates of: small for gestational age (<10th and <3rd percentiles)
Neonatal morbidity (NICU) | Throughout pregnancy until 6-12 weeks postpartum
  Rates of: neonatal ICU admission
Neonatal morbidity (apgar) | Throughout pregnancy until 6-12 weeks postpartum
  Rates of: low Apgar (<4 at 5 min)
Fetal and neonatal morbidity | Throughout pregnancy until 6-12 weeks postpartum
  Rates of: stillbirth, spontaneous abortion, elective termination
Maternal morbidity | Throughout pregnancy until 6-12 weeks postpartum
  Rates of: gestational diabetes, pre-eclampsia, placental abruption
Mode of delivery | Through study completion, about every 9-months
  Rates of cesarean sections and vaginal deliveries
Child growth (weight) | 6-12 weeks postpartum
  weight
Child growth (head circumference) | 6-12 weeks postpartum
  head circumference
Child growth (height) | 6-12 weeks postpartum
  length
Child Major Illnesses/conditions | Delivery to 6-12 weeks postpartum
  Proportion of children receiving diagnoses of major illness/conditions
Hospitalizations | Delivery to 6-12 weeks postpartum
  Proportion of mothers and infants re-admitted to hospital
Emergency care visits | Delivery to 6-12 weeks postpartum
  Proportion of mothers and infants with emergency care visits

CONTACTS AND LOCATIONS:
Overall Officials: Mark Walker, MD, MSc, MHM, Principal Investigator — Ottawa Hospital Research Institute; Daniel Corsi, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramlawi S, Murphy MSQ, Dingwall-Harvey ALJ, Rennicks White R, Gaudet LM, McGee A, DeGrace A, Cantin C, El-Chaar D, Walker MC, Corsi DJ. Cannabis Use in Pregnancy and Downstream effects on maternal and infant health (CUPiD): a protocol for a birth cohort pilot study. BMJ Open. 2022 Dec 22;12(12):e066196. doi: 10.1136/bmjopen-2022-066196. PMID 36549747